CLINICAL TRIAL: NCT03461146
Title: A Phase III, Open-label Study of MT-6548 in Hemodialysis Subjects With Anemia Associated With Chronic Kidney Disease in Japan
Brief Title: Efficacy and Safety Study to Evaluate MT-6548 in Hemodialysis Subjects Not Receiving ESAs With Anemia Associated With Chronic Kidney Disease in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-6548-J04
Record Dates: First submitted 2018-03-05; First posted 2018-03-09 (Actual); Results first posted 2021-05-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Anemia; Hemodialysis Dependent Chronic Kidney Disease
MeSH Terms: conditions — Anemia | interventions — vadadustat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MT-6548 (Experimental)
  Interventions: Drug: MT-6548

INTERVENTIONS:
Drug: MT-6548 — Oral tablet
  Other Names: vadadustat; AKB-6548

SUMMARY:
For hemodialysis subjects not receiving ESAs with anemia associated with chronic kidney disease, evaluate Hb correction and maintenance effect and safety of MT-6548.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CKD
* Receiving hemodialysis or hemodiafiltration 3 times a week for more than 12 weeks prior to the screening period, excluding receiving home dialysis or combination of peritoneal dialysis.
* Not being treated with ESAs or if being treated with ESAs, leave defined interval between last ESAs administration and the first day of the screening period
* Mean of the two screening Hb levels closest in time to the baseline visit is ≥8.0 g/dL and <10.0 g/dL
* Fluctuation between the two Hb levels closest in time to the baseline visit during the screening period less than 1.5 g/dL
* Serum ferritin ≥ 100 ng/mL, or TSAT ≥20% during the screening period
* Folate and vitamin B12 ≥ lower limit of normal during the screening period

Exclusion Criteria:

* Anemia due to a main cause other than CKD: sickle cell disease, myelodysplastic syndrome, bone marrow fibrosis, hematologic malignancy, hemolytic anemia, thalassemia, or pure red cell aplasia
* Active bleeding or recent blood loss within 8 weeks prior to the screening period
* RBC transfusion within 8 weeks prior to the screening period
* Received testosterone enanthate or mepitiostane within 8 weeks prior to the screening period
* AST, ALT, or total bilirubin >2.5 x upper limit of normal during the screening period
* Uncontrolled hypertension (diastolic blood pressure >110 mm Hg or systolic blood pressure >180 mm Hg) at the first day of the screening period and Day 1
* Ophthalmic examinations during the screening period correspond to either of the following criteria;

  * No available fundal findings
  * Findings indicating the presence of active fundal disease
* Severe heart failure (New York Heart Association Class IV)
* Cerebrovascular disorder or acute coronary syndrome (hospitalization due to unstable angina or myocardial infarction), requiring hospitalization due to urgent percutaneous intervention for coronary or heart failure within 12 weeks prior to the screening period
* Current or history of malignancy. History of malignancy with no recurrence for the recent 5 years is not an exclusion criterion
* New onset or recurrent event of deep vein thrombosis or pulmonary embolism within 12 weeks prior to the screening period
* Current or history of hemosiderosis or hemochromatosis
* History of prior organ transplantation or scheduled organ transplant, or prior transplantation of hematopoietic stem cell or bone marrow
* Males and females of childbearing potential who are unwilling to use an acceptable method of contraception during the designated period (Males: during the study and 90 days after the last dose, females: during study and 30 days after the last dose)
* Females who are pregnant or breast feeding, or are predicted to be pregnant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (16):
- Japan (16):
  - Research site, Aichi
  - Research site, Chiba
  - Research site, Fukushima
  - Research site, Gunma
  - Research site, Hokkaido
  - Research site, Hyōgo
  - Research site, Ibaraki
  - Research site, Kagoshima
  - Research site, Nagano
  - Research site, Okayama
  - Research site, Okinawa
  - Research site, Osaka
  - Research site, Saitama
  - Research site, Shiga
  - Research site, Shizuoka
  - Research site, Yamagata

REFERENCES:
- [Result] Nangaku M, Kondo K, Takabe S, Ueta K, Tandai T, Kawaguchi Y, Komatsu Y. A phase 3, open-label, single-arm study of vadadustat for anemia in chronic kidney disease for Japanese patients on hemodialysis not receiving erythropoiesis-stimulating agents. Ther Apher Dial. 2022 Feb;26(1):45-54. doi: 10.1111/1744-9987.13699. Epub 2021 Jun 28. PMID 34115437

RESULTS

PARTICIPANT FLOW:
Groups:
- MT-6548: MT-6548: Oral tablet. The dose was adjusted to 150-600 mg/day according to the pre-specified dose adjustment algorithm.
Period: Overall Study
Arm/Group | MT-6548
Started | 24
Completed | 21
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | MT-6548
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian (Japanese) | 24
  Asian (Other) | 0
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Hb Level of Week 20 and Week 24
Time Frame: Up to Week 24
Population: This analysis was performed in subjects who measured Hb at least one visit after baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | MT-6548
Number analyzed (Participants) | 23
g/dL | 10.75 [10.35 to 11.14]

2. Primary Outcome: Hb Level at Each Assessment Time Point
Time Frame: Up to Week 24
Population: This analysis was performed only in subjects who have Hb data at each visit.
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | MT-6548
Number analyzed (Participants) | 24
g/dL
  Baseline | 9.15 [8.73 to 9.57]
  Week 2: number analyzed (Participants) | 23
  Week 2 | 9.25 [8.83 to 9.68]
  Week 4: number analyzed (Participants) | 22
  Week 4 | 9.53 [9.03 to 10.04]
  Week 6: number analyzed (Participants) | 21
  Week 6 | 9.90 [9.37 to 10.43]
  Week 8: number analyzed (Participants) | 20
  Week 8 | 10.33 [9.80 to 10.85]
  Week 10: number analyzed (Participants) | 19
  Week 10 | 10.56 [10.08 to 11.04]
  Week 12: number analyzed (Participants) | 19
  Week 12 | 10.68 [10.18 to 11.19]
  Week 16: number analyzed (Participants) | 19
  Week 16 | 11.17 [10.66 to 11.68]
  Week 20: number analyzed (Participants) | 19
  Week 20 | 11.08 [10.73 to 11.43]
  Week 24: number analyzed (Participants) | 19
  Week 24 | 11.03 [10.60 to 11.45]
  Week 24 (LOCF): number analyzed (Participants) | 23
  Week 24 (LOCF) | 10.56 [9.95 to 11.17]

3. Primary Outcome: Percentage of Subjects With Hb Level at Each Assessment Time Point Within the Target Range During the Treatment Period
Time Frame: Up to Week 24
Population: This analysis was performed only in subjects who have Hb data at each visit.
Measure: Number; unit: percentage of subjects
Arm/Group | MT-6548
Number analyzed (Participants) | 24
percentage of subjects
  Baseline | 16.7
  Week 2: number analyzed (Participants) | 23
  Week 2 | 21.7
  Week 4: number analyzed (Participants) | 22
  Week 4 | 36.4
  Week 6: number analyzed (Participants) | 21
  Week 6 | 47.6
  Week 8: number analyzed (Participants) | 20
  Week 8 | 55.0
  Week 10: number analyzed (Participants) | 19
  Week 10 | 63.2
  Week 12: number analyzed (Participants) | 19
  Week 12 | 68.4
  Week 16: number analyzed (Participants) | 19
  Week 16 | 63.2
  Week 20: number analyzed (Participants) | 19
  Week 20 | 78.9
  Week 24: number analyzed (Participants) | 19
  Week 24 | 73.7

4. Primary Outcome: Time to Reach the Target Hb Range
Time Frame: Up to Week 24
Population: This analysis was performed except for subjects with Hb of 10.0 g/dL or more at baseline.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | MT-6548
Number analyzed (Participants) | 20
days | 67.2 [45.8 to 88.6]

5. Primary Outcome: Rate of Increase in Hb Level
Time Frame: Up to Week 6
Population: This analysis was performed in subjects who measured Hb up to week 4 or week 6.
Measure: Mean (95% Confidence Interval); unit: g/dL/week
Arm/Group | MT-6548
Number analyzed (Participants) | 22
g/dL/week
  Calculated based on Hb at baseline and Week 4 | 0.05 [-0.05 to 0.16]
  Calculated based on Hb up to Week6: number analyzed (Participants) | 21
  Calculated based on Hb up to Week6 | 0.09 [0.01 to 0.17]

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | MT-6548
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 7/24
Other Adverse Events (participants affected / at risk) | 15/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MT-6548 (N=24)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Shunt stenosis (Injury, poisoning and procedural complications) | 1
Vascular access malfunction (Injury, poisoning and procedural complications) | 1
Aneurysm (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MT-6548 (N=24)
Diarrhoea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Nasopharyngitis (Infections and infestations) | 5
Shunt stenosis (Injury, poisoning and procedural complications) | 5
Skin abrasion (Injury, poisoning and procedural complications) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-12-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT03461146/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT03461146/SAP_001.pdf